CLINICAL TRIAL: NCT03591848
Title: Evaluation of an Online Decision Support Tool for Young Women With Breast Cancer During the Proposal for Preservation of Fertility
Brief Title: Pilot Study of a Web-based Decision Aid for Young Women With Breast Cancer, During the Proposal for Preservation of Fertility
Acronym: DECISIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: K171005J; 2017-A03008-45 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Preservation of fertility; Online support decision tool
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DECISIF (Experimental): Exposed to an online support decision tool, in addition of the standard oral information
  Interventions: Behavioral: Online support decision tool; Behavioral: standard oral information
- IRIS (Active Comparator): Exposed to a standard oral information
  Interventions: Behavioral: standard oral information

INTERVENTIONS:
Behavioral: Online support decision tool — Online support decision tool, in addition of the standard oral information
  Arms: DECISIF
Behavioral: standard oral information — standard oral information

SUMMARY:
Comparative study of two information modalities during the care course, aiming to propose the preservation of fertility to young women with breast cancer (but not yet under treatment): standard oral information during the PF consultation vs. an online decision support tool, consulted prior to the PF consultation, during which the standard oral information is provided.

DETAILED DESCRIPTION:
In recent decades, the incidence of breast cancer has increased significantly among young women. Between 1980 and 2012, there was an increase of 59% and 53% in the 30-39 age group and the 40-49 age group, respectively. However, both diagnostic and therapeutic advances made it possible to significantly reduce mortality, at the cost of potentially deleterious chemotherapeutic treatments for reproductive function. These treatments may therefore be the cause of a chronic pathology "infertility" that may negatively impact the quality of life of young breast cancer survivors.

Since 2004, in France, the preservation of fertility (PF) is part of the different laws of bioethics. The latest cancer plans have highlighted the importance of quality of life in patients cured of cancer. For young women, this often involves the possibility of accessing maternity, using their own gametes. Thus, access to an onco fertility consultation should be systematically proposed, ideally before the initiation of any cancer treatment.

While the importance of oncofertility consultations is now recognized, they raise a certain number of ethical questions, particularly as to the nature of the information to be transmitted, whether it is generalizable or not, and how it is delivered and supported.

Very little data on the value of decision support tools in PF for women with breast cancer are available, while the concept of "shared medical decision" is becoming increasingly important in the doctor-patient relationship.

The only available studies have shown that these tools can reduce the level of decisional conflict and regret over fertility-related treatment options, and improve knowledge about fertility and satisfaction among young women.

This study aims to compare two modalities of delivery of information to breast cancer patients (not yet under treatment): standard oral information during the prevention of fertility (PF) consultation vs. an online decision support tool, consulted prior to the PF consultation, during which the standard oral information is provided.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years women
* with breast cancer
* cancer treatment not started, no antecedent of chemotherapy
* speaking French
* affiliated in Social Insurance

Exclusion Criteria:

* recurrence of breast cancer
* metastatic breast cancer
* pregnancy in progress
* Adults protected (wardship, guardianship, protection of justice)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 186 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Multidimensional Measure of Informed Choice (MMIC) | 1 day (During the PF consultation)
  Measure of patient autonomy for making decision, according to the Multidimensional Measure of Informed Choice (MMIC).
  A series of closed questions (based on the Osgoog's scale) on their feelings about this fertility preservation approach, describing attitudes in regards to "good / bad", "important / unimportant", "unhelpful" good thing / bad thing, "" pleasant / unpleasant "and" useful / useless ". Responses go from "very positive" (1) to "very negative" (7).

SECONDARY OUTCOMES:
Decisional Conflict Scale Measure on | 1 day (at the end of the PF consultation)
  patient's decision-making discomfort, specific support needs for decision-making, the quality of decision making, the impact of supportive interventions on health decision-making.
Anxiety | 1 day ( at the end of the PF consultation)
  : the 6 items of State and Trait Anxiety Inventory [55] [56], a reliable and sensitive measure of anxiety will be used to assess emotional disturbance. It consists of 6 items, indicating the lowest level of anxiety (1 = not at all) and 4 the highest (4 = very much), with a reverse rating items. The items are summated multiplied by 20 and divided by 6. Patients with scores> 50 are considered to have a high level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Michaël GRYNBERG, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Reproduction medicine and fertility preservation ANTOINE BECLERE Hospital, Clamart, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benoit A, Grynberg M, Morello R, Sermondade N, Grandazzi G, Moutel G. Does a web-based decision aid improve informed choice for fertility preservation in women with breast cancer (DECISIF)? Study protocol for a randomised controlled trial. BMJ Open. 2020 Feb 10;10(2):e031739. doi: 10.1136/bmjopen-2019-031739. PMID 32047010